CLINICAL TRIAL: NCT01488045
Title: Randomized Trial to Compare Propofol to Fentanyl and Midazolam for Colonoscopy.
Brief Title: Compare Propofol to Fentanyl and Midazolam for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCCS 262
Record Dates: First submitted 2011-12-01; First posted 2011-12-08 (Estimated); Results first posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Colon Cancer; Rectal Cancer; Colonic Diverticulosis
Keywords: Colonoscopy; Propofol; Cancer Screening
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Diverticulosis, Colonic | interventions — Fentanyl; Propofol; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl and Midazolam (Active Comparator): Fentanyl and Midazolam sedation for colonoscopy discomfort
  Interventions: Drug: Fentanyl; Drug: Midazolam
- Propofol (Active Comparator): Propofol sedation for colonoscopy discomfort
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Fentanyl — Fentanyl will be administered IV according to standard procedure for colonoscopy. Initial dose will consist of no more than 50µg of Fentanyl. Patient response will be monitored for 30-60 seconds of observation before deciding to administer more Fentanyl in no more than 50µg increments. increments.
  Other Names: Durogesic; Duragesic; Matrifen
  Arms: Fentanyl and Midazolam
Drug: Propofol — Propofol will be administered IV according to standard procedure for colonoscopy. The initial bolus of propofol will be up to 60 mg IV. Patient response will be monitored for 30-60 seconds of observation before deciding to administer more sedation in 10-20 mg boluses.
  Other Names: Diprivan
  Arms: Propofol
Drug: Midazolam — Midazolam will be administered IV according to standard procedure for colonoscopy. Initial dose will consist of no more than 2 mg of Midazolam. Patient response will be monitored for 30-60 seconds of observation before deciding to administer more Midazolam in no more than 2 mg increments.
  Other Names: Versed
  Arms: Fentanyl and Midazolam

SUMMARY:
The study aim is to determine if Propofol or the combination of Fentanyl and low-dose Midazolam, are equivalent for patient satisfaction and discomfort when undergoing a colonoscopy. This is a prospective randomized study of 262. The primary outcome of this study is participant's satisfaction and discomfort of the colonoscopy procedure as perceived by the participant, and the secondary outcome will be the discomfort of the patient and difficulty of the procedure as perceived by the physician.

DETAILED DESCRIPTION:
Background The use of colonoscopy has become an important diagnostic and therapeutic tool in the evaluation of multiple medical conditions of the gastrointestinal tract. Despite its widespread use, there continues to be debate concerning the best pharmacologic approach to patient satisfaction and discomfort of the procedure and to minimize side effects.

Aim Two standard pharmacologic (Propofol or Fentanyl and low-dose Midazolam) approaches for colonoscopy will be evaluated systematically to determine if these two approaches are equivalent in terms of patient rating of satisfaction and patient discomfort to the procedure and side effects

Study Design This is a prospective randomized study of 262 participants undergoing outpatient colonoscopy at an independent academic medical center. The primary outcome of this study is participant's satisfaction, and the secondary outcome is discomfort of the patient as perceived by the physician performing the procedure.

Other Variables of Interest.

* Duration of procedure as defined by time the patient arrives in the room to the time the patient is appropriate for discharge.
* Difficulty of procedure rated by the physician on a scale of 0-10
* Colonoscopy completion rates (intubation of cecum).
* Complications including oxygen desaturation or hypotension.
* Cost of the two medication regiments

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Elective outpatient colonoscopy
* American Society of Anesthesiology Class (ASA) < IV

Exclusion Criteria:

* Age < 18
* Inpatient status
* Emergency procedure
* History of colonic or rectal resection
* History of hypersensitivity to Propofol (or soy or egg products),Fentanyl or Midazolam
* ASA of IV
* Neurological deficit
* Acute gastrointestinal bleeding
* On anticoagulation agents
* Noncompliance with bowel regiment
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2011-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cleary, MD, Principal Investigator — Trinity Health Michigan
Locations (1):
- Saint Joseph Mercy Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- See also: American Society of Colon and Rectal Surgeons — http://www.fascrs.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fentanyl and Midazolam | Propofol
Started | 145 (Approved by IRB 3/11/11 Enrollment start date) | 144 (3/11/2011 Approved by IRB and enrollment started.)
Completed | 136 (Enrollment target number met on 10/10/14) | 126 (Target number met on 10/10/14)
Not Completed | 9 | 18
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Failure to present for colonoscopy | 3 | 6
Not completed — Failure to report exclusion criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Propofol Intervention: Propofol: an initial dose of ≤60 mg intravenously, with additional dosing at the discretion of the anesthesia provider.
- Midazolam/Fentanyl Intervention: Fentanyl: Fentanyl will be administered IV according to standard procedure for colonoscopy. Initial dose will consist of no more than 50µg of Fentanyl. Patient response will be monitored for 30-60 seconds of observation before deciding to administer more Fentanyl in no more than 50µg increments. increments.
  Midazolam: Midazolam will be administered IV according to standard procedure for colonoscopy. Initial dose will consist of no more than 2 mg of Midazolam. Patient response will be monitored for 30-60 seconds of observation before deciding to administer more Midazolam in no more than 2 mg increments.
- Total: Total of all reporting groups
Arm/Group | Propofol Intervention | Midazolam/Fentanyl Intervention | Total
Number analyzed (Participants) | 126 | 136 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (13.4) | 58.1 (13.8) | 57.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 60 | 121
  Male | 65 | 76 | 141
BMI >=30 [Count of Participants; unit: Participants] — Body Mass Index is an index calculated by a person's weight in kilograms divided by the square of height in meters. In this case, the study used a categorical variable of BMI greater than or equal to 30 (yes, no)
  Participants | 38 | 41 | 79
General health factors [Count of Participants; unit: Participants] — Comorbidities present at surgery
  Participants
    Congestive heart failure | 1 | 1 | 2
    History of myocardial infarction | 2 | 4 | 6
    Diabetes mellitus | 8 | 10 | 18
    Chronic obstructive pulmonary disease | 2 | 5 | 7
    Obstructive sleep apnea | 10 | 12 | 22
    History of diverticulitis | 5 | 8 | 13
    IBD | 1 | 2 | 3
    Ongoing malignancy | 3 | 2 | 5
Procedure/recovery times (min) [Mean (Standard Deviation); unit: minutes]
  Procedure time | 23.0 (9.1) | 24.4 (9.3) | 23.73 (9.23)
  Recovery time | 35.0 (7.3) | 33.6 (15.0) | 34.27 (11.95)
  Time in colonoscopy suite | 34.4 (10.3) | 38.7 (9.7) | 36.63 (10.22)
Amount of anesthetic drug used [Mean (Standard Deviation); unit: units] — Population: The Row population represents the patients who received that drug which is specific to each Intervention Arm. The Propofol patient group would only receive Propofol (no Midazolam/Fentanyl received), and the M/F group would only receive Midazolam and Fentanyl (no propofol).
  units
    Midazolam, mg: number analyzed (Participants) | 0 | 136 | 136
    Midazolam, mg |  | 5.7 (1.4) | 5.7 (1.4)
    Fentanyl, μg: number analyzed (Participants) | 0 | 136 | 136
    Fentanyl, μg |  | 138.8 (41.6) | 138.8 (41.6)
    Propofol, mg: number analyzed (Participants) | 126 | 0 | 126
    Propofol, mg | 341.0 (122.8) |  | 341.0 (122.8)
Cecum intubation [Count of Participants; unit: Participants] — Categorical variable
  Participants | 111 | 116 | 227

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction Scores (Absolute Value)
Description: Measured by the patient using a 100-point Visual Analog Scale (VAS) [0-100%] with higher score indicating higher agreement with the statement/question. Higher agreement scores would indicate higher satisfaction (better outcome).
Time Frame: Survey administered in the recovery room up to 30 minutes following procedure ("Recovery room"), and a follow-up patient survey was carried out by telephone between 1 and 5 days postprocedure ("1-5 d postprocedure")
Population: All patients who completed the intervention were included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propofol Intervention | Midazolam/Fentanyl Intervention
Number analyzed (Participants) | 126 | 136
score on a scale
  Recovery Room: Satisfaction with colonoscopy | 98.0 (12.8) | 83.9 (28.3)
  Recovery Room: Would undergo another colonoscopy with same sedation | 98.1 (12.6) | 79.2 (36.0)
  Recovery Room: Would encourage others to have same sedation | 100.0 (0) | 79.5 (37.9)
  Recovery Room: Comfort | 88.8 (25.5) | 86.1 (25.0)
  1-5 d postprocedure: Satisfaction with colonoscopy | 98.7 (9.4) | 79.8 (34.1)
  1-5d postprocedure: Would undergo another colonoscopy with same sedation | 98.2 (12.9) | 73.9 (41.4)
  1-5d postprocedure: Would encourage others to have same sedation | 98.2 (13.0) | 74.5 (41.2)
  1-5d postprocedure: Comfort | 94.7 (16.5) | 84.4 (28.9)
Statistical Analysis 1: Comparison: Propofol Intervention vs Midazolam/Fentanyl Intervention; To calculate the required sample size for this study, the equivalence limit was set at 5 units difference on the VAS, with an expected mean difference of 0. The common SD of 16.2 was estimated based on the range of expected scores for the VAS from Ulmer et al. Using these inputs, a total sample size of 262 patients was estimated to have 80% power to reject the null hypothesis that the test and standard were not equivalent and conclude that they were equivalent; Test type: Equivalence — We compared patient satisfaction for those receiving the 2 sedation regimens using the Schuirmann 2 one-sided t test procedure.15 The groups were declared to be equivalent in terms of patient satisfaction if the 90% CI for the difference in mean satisfaction had outer boundaries indicating <5% difference on the 100-point VAS. Nonequivalence was declared if the lower 90% CI boundary for the difference was less than -5.0, or if the upper 90% CI boundary for the difference was >5.0; Mean Difference (Final Values) = -14.0741, 95% CI 2-sided [-18.5 to -9.6], Standard Deviation 22.2

2. Secondary Outcome: Patient Pain & Discomfort Rating (Absolute Value)
Description: Self-reported by patient via a Visual Analog Scale [0-10], where 0=no pain, 10=worst possible pain
Time Frame: as for outcome 1
Population: All patients who completed the intervention were included
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propofol Intervention | Midazolam/Fentanyl Intervention
Number analyzed (Participants) | 126 | 136
score on a scale
  Recovery room: patient highest pain | 0.2 (0.9) | 2.4 (3.1)
  Recovery room: Average pain | 0.8 (0.4) | 1.9 (2.6)
  Recovery room: Average discomfort during recovery | 0.7 (1.7) | 1.2 (2.1)
  1-5d postprocedure: Highest pain | 0.16 (1.0) | 1.9 (3.2)
  1-5d postprocedure: Average pain | 0.4 (1.4) | 0.7 (2.0)
  1-5d postprocedure: Average discomfort during recovery | 0.17 (1.0) | 1.7 (3.0)

3. Secondary Outcome: Physician Perceptions (Absolute Value)
Description: Self-reported Physician/Endoscopist perceptions Measured via Visual Analog Scale [0-10] of: Highest pain, Average pain, Difficulty of procedure, Bowel preparation, Patient movement. A score of 0 on the scale=no pain/difficulty, while a score of 10=worst possible pain/difficulty/severity. The higher the score the worse the outcome.
Time Frame: Measured via physician survey within 30 minutes after the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propofol Intervention | Midazolam/Fentanyl Intervention
Number analyzed (Participants) | 126 | 136
score on a scale
  Endoscopist rating: Highest Pain | 1.3 (1.8) | 3.7 (2.4)
  Endoscopist rating: Average Pain | 0.6 (0.8) | 2.1 (1.8)
  Endoscopist rating: Difficulty of Procedure | 4.4 (2.7) | 5.2 (2.5)
  Endoscopist rating: Bowel preparation | 1.4 (0.6) | 1.3 (0.6)
  Endoscopist rating: Patient Movement | 1.3 (2.2) | 1.6 (1.7)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the procedure and while the patient was in recovery, (the time the patient was in the OR to the time patient had recovered, up to 30 minutes).
Arm/Group | Propofol Intervention | Midazolam/Fentanyl Intervention
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/136
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/136
Other Adverse Events (participants affected / at risk) | 18/126 | 19/136
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Propofol Intervention (N=126) | Midazolam/Fentanyl Intervention (N=136)
Decreased oxygen saturation (Surgical and medical procedures) | 6 | 13
Decreased heart rate (Surgical and medical procedures) | 6 | 2
Decreased blood pressure (Surgical and medical procedures) | 3 | 2
Airway intervention (Surgical and medical procedures) | 3 | 2
Mechanical ventilation (Surgical and medical procedures) | 0 | 0

LIMITATIONS AND CAVEATS:
This is a single-institution, single endoscopist study and is limited by the inability to perform blinding of the endoscopist.The endoscopist could not be blinded to treatment because of the presence of an anesthesia provider in the colonoscopy suite for the Propofol group. Anesthesia providers were not present for the midazolam/fentanyl group because we wanted to mimic and compare 2 of the most commonly used practice strategies as much as possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes